CLINICAL TRIAL: NCT00480272
Title: A Phase IV Multicenter, Randomized, Double-blind Study. prospeCtive Study on Intensive Early Rheumatoid Arthritis Treatment With adalimUmab: Induction of REmission and Maintenance
Brief Title: Prospective Study on Intensive Early Rheumatoid Arthritis Treatment
Acronym: CURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carlomaurizio Montecucco, Director, Academic Division of Rheumatology, IRCCS Policlinico S. Matteo and University of Pavia, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CURE; 2006-003843-22 (EudraCT Number)
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; clinical remission
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; deltacortene; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Experimental): * adalimumab 40 mg subcutaneous injections every other week from baseline to month 12
  * methotrexate orally weekly at initial dose of 10 mg rising to 20 mg weekly over 4 weeks in 2.5 mg increments, continued up to month 24.
  * prednisone orally 50 mg daily, gradually tapered up to 6.25 mg at week 7 and stopped at month 6
  Interventions: Drug: adalimumab, plus prednisone
- group B (Placebo Comparator): * adalimumab 40 mg subcutaneous injections every other week from baseline to the end of month 12
  * methotrexate orally oweekly at an initial dose of 10 mg rising to 20 mg weekly over 4 weeks in 2.5 mg increments, continued up to month 24.
  * placebo orally, stopped at month 6
  Interventions: Drug: adalimumab plus placebo

INTERVENTIONS:
Drug: adalimumab, plus prednisone — adalimumab 40 mg/sc every 2 weeks plus methotrexate 20 mg/po every week plus placebo or prednisone 50 mg/po day then reduced to 6.25/po day
  Other Names: humira (adalimumab); deltacortene (prednisone)
  Arms: group A
Drug: adalimumab plus placebo — adalimumab 40 mg/sc every 2 weeks plus methotrexate 20 mg/po every week plus placebo daily for 6 months
  Other Names: humira (adalimumab)
  Arms: group B

SUMMARY:
Hypothesis: Early intensive treatment with anti-TNF agent plus methotrexate plus high dose prednisone may increase remission rate and may induce stable remission in Rheumatoid Arthritis Objective: to evaluate induction of remission using adalimumab, prednisone and methotrexate and maintenance of remission after discontinuation of adalimumab and prednisone

DETAILED DESCRIPTION:
Treatment group A 0 - 6 months: Adalimumab 40 mg eow + methotrexate rapidly titrated to 20 mg weekly + prednisone 50 mg/d tapered to 6.25 mg 6 - 12 months: Adalimumab 40 mg eow plus methotrexate 20 mg weekly group B 0 - 6 months: Adalimumab 40 mg eow + methotrexate rapidly titrated to 20 mg weekly + placebo 6 - 12 months: Adalimumab 40 mg eow + methotrexate rapidly titrated to 20 mg weekly

Follow up period - Open Label phase:

Patients achieving clinical remission will be than treated only with MTX and observed for another 12 months period. Patients who do not achieve clinical remission or patients who will experience a relapse of the disease will be treated according to standard of care (SOC) modalities.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis diagnosed for at least 6 weeks, but no more than 1 year, according to the revised 1987 ACR criteria
* Naïve to treatment with MTX
* Swollen joint count (SJC) > 8 tender joint count (TJC) > 8
* At screening CRP > 1.5 mg/dL (15 mg/L) or ESR ≥ 28 mm/h
* ≥ 1 joint erosion or RF positivity or anti-CCP positivity
* Age 18-70 years.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* Functional class IV
* Any surgical procedure within 12 weeks prior to baseline or planned during the study.
* Pregnancy or breast feeding.
* Evidence of significant concomitant disease
* Primary or secondary immunodeficiency
* active infection of any kind
* History of previously untreated infection with mycobacterium tuberculosis or current treatment for same.
* History of cancer
* Any history or presence of congestive heart failure (CHF) (New York Heart Association classification for CHF: Class III or IV).
* Any history of myocardial infarction within 5 years.
* History of a severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of adalimumab or methotrexate.
* Positive serology for hepatitis B or C indicating active infection.
* Hemoglobin < 8.0 g/dL.
* Absolute neutrophil count (ANC) < 1.5 x 103/L.
* Liver function abnormality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2007-05; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the proportion of subjects who achieve remission at week 52 after treatment, as defined by DAS 28 </= 2.6 | 52 weeks

SECONDARY OUTCOMES:
subjects who maintain stable remission at 24 months; ACR 20,50,70 at month 4,8,12,24; DAS 28 at month 4,8,12,24; HAQ at week 0,4,8,12,24; radiographic progression at months 12, 24; safety of different treatment regimens | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: carlomaurizio montecucco, MD, Principal Investigator — IRCCS S. Matteo Foundation, Pavia
Locations (1):
- IRCCS S. Matteo Hospital, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No